CLINICAL TRIAL: NCT02643004
Title: The Clinical Comparison of Senofilcon A and Stenfilcon A Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-62
Record Dates: First submitted 2015-12-28; First posted 2015-12-30 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Senofilcon A (Active Comparator): Participants were randomized to wear senofilcon A lens pair for one week during the crossover study.
  Interventions: Device: Senofilcon A
- Stenfilcon A (Active Comparator): Participants were randomized to wear stenfilcon A lens pair for one week during the crossover study.
  Interventions: Device: Stenfilcon A

INTERVENTIONS:
Device: Senofilcon A — contact lens
  Arms: Senofilcon A
Device: Stenfilcon A — contact lens
  Arms: Stenfilcon A

SUMMARY:
The objective of this study is to compare the clinical performance of senofilcon A lens with the stenfilcon A lens each for one week of daily disposable wear.

DETAILED DESCRIPTION:
The purpose of this bilateral cross-over study is to evaluate the clinical performance of senofilcon A lens with the stenfilcon A lens. In particular, the study will focus on ocular physiology, lens fit, lens surface, visual acuity, and subjective response.

ELIGIBILITY:
Inclusion criteria

Subjects will only be eligible for the study if:

* They are of legal age (18) and capacity to volunteer.
* They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
* They are willing and able to follow the protocol.
* They agree not to participate in other clinical research for the duration of this study.
* They have a contact lens spherical prescription between -1.00 to - 6.00D (inclusive)
* They have a spectacle cylindrical correction of -0.75D or less in each eye.
* At dispensing, they can attain at least 0.10 logMAR distance high contrast visual acuity in each eye with the study lenses within the available power range.
* They currently use soft contact lenses or have done so in the previous six months.
* They are willing to comply with the wear schedule (at least six days per week and for at least eight hours per day).

Exclusion criteria

Subjects will not be eligible to take part in the study if:

* They have an ocular disorder which would normally contra-indicate contact lens wear.
* They have a systemic disorder which would normally contra-indicate contact lens wear.
* They are using any topical medication such as eye drops or ointment.
* They have had cataract surgery.
* They have had corneal refractive surgery.
* They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
* They are pregnant or lactating.
* They have any ocular abnormality which would, in the opinion of the investigator, normally contraindicate contact lens wear.
* They have any infectious disease which would, in the opinion of the investigator, contraindicate contact lens wear or pose a risk to study personnel; or they have any immunosuppressive disease (e.g. HIV), or a history of anaphylaxis or severe allergic reaction.
* They have taken part in any other contact lens or care solution clinical trial or research, within two weeks prior to starting this study.
* They currently wear either MyDay (daily) or the Acuvue Oasys (2 weekly) lens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carole Maldonado-Codinal, PhD, Principal Investigator — Eurolens Research, University of Manchester
Locations (1):
- Eurolens Research - The University of Manchester, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Senofilcon A, Then Stenfilcon A: Participants were randomized to wear senofilcon A lens pair for one week during the crossover study.
  Senofilcon A: contact lens
  Stenfilcon A: contact lens
- Stenfilcon A, Then Senofilcon A: Participants were randomized to wear stenfilcon A lens pair for one week during the crossover study.
  Stenfilcon A: contact lens
  Senofilcon A: contact lens
Period: First Intervention (One Week)
Arm/Group | Senofilcon A, Then Stenfilcon A | Stenfilcon A, Then Senofilcon A
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0
Period: Second Intervention (One Week)
Arm/Group | Senofilcon A, Then Stenfilcon A | Stenfilcon A, Then Senofilcon A
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Baseline Characteristics: Participants were randomized to wear senofilcon A or stenfilcon A lens pair for one week during the crossover study.
  Senofilcon A: contact lens
  Stenfilcon A: contact lens
Arm/Group | Overall Baseline Characteristics
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Ocular Physiology
Description: Ocular physiology assessment of senofilcon A and stenfilcon A lenses by biomicroscopy for the following: corneal staining, conjunctival hyperaemia, limbal hyperaemia, and conjunctival staining. Scale 0-4, 0.25 steps, 0=normal, 4=severe.
Time Frame: Baseline and 1 week
Population: Protocol deviations occurred for 2 participants and therefore resulted in incomplete data sets.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 70 | 70
units on a scale
  Baseline - Corneal staining | 0.13 (0.30) | 0.13 (0.30)
  1 week - Corneal staining: number analyzed (Participants) | 70 | 69
  1 week - Corneal staining | 0.21 (0.34) | 0.15 (0.29)
  Baseline - Conjunctival staining | 0.21 (0.30) | 0.21 (0.30)
  1 week - Conjunctival staining: number analyzed (Participants) | 70 | 69
  1 week - Conjunctival staining | 0.82 (0.51) | 0.48 (0.43)
  Baseline - Conjunctival hyperaemia | 0.81 (0.23) | 0.81 (0.23)
  1 week - Conjunctival hyperaemia: number analyzed (Participants) | 69 | 70
  1 week - Conjunctival hyperaemia | 0.82 (0.25) | 0.86 (0.24)
  Baseline - Limbal hyperaemia | 0.70 (0.28) | 0.70 (0.28)
  1 week - Limbal hyperaemia: number analyzed (Participants) | 69 | 68
  1 week - Limbal hyperaemia | 0.69 (0.26) | 0.75 (0.26)

2. Primary Outcome: Overall Subjective Score of Lenses
Description: Subjective responses will be evaluated for each pair using questionnaire. Scale 0-100, 0=extremely poor, 100=excellent.
Time Frame: Baseline and 1 week
Population: A protocol deviation occurred for 1 participant and therefore resulted in incomplete data sets.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 70 | 70
units on a scale
  Baseline | 92.3 (8.8) | 89.4 (11.1)
  1 week: number analyzed (Participants) | 70 | 69
  1 week | 87.0 (13.1) | 80.0 (18.3)

3. Primary Outcome: Comfort
Description: Subjective responses for comfort will be evaluated for each pair using questionnaire. Scale 0-100, 0=causes pain, cannot be tolerated, 100=excellent, cannot be felt.
Time Frame: Baseline and 1 week
Population: A protocol deviation occurred for 1 participant and therefore resulted in incomplete data sets.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 70 | 70
units on a scale
  Baseline | 90.8 (10.2) | 90.5 (10.7)
  1 week: number analyzed (Participants) | 70 | 69
  1 week | 87.0 (11.5) | 82.1 (14.0)

4. Primary Outcome: Dryness
Description: Subjective responses for dryness will be evaluated for each pair using questionnaire. Scale 0-100, 0=extremely poor, high levels of dryness, 100=excellent, no dryness.
Time Frame: 1 week
Population: A protocol deviation occurred for 1 participant and therefore resulted in incomplete data sets.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 70 | 69
units on a scale | 82.3 (14.3) | 77.7 (17.8)

5. Primary Outcome: Vision
Description: Subjective responses for vision will be evaluated for each pair using questionnaire. Scale 0-100, 0=unacceptable, lens cannot be worn, 100=excellent.
Time Frame: Baseline and 1 week
Population: A protocol deviation occurred for 1 participant and therefore resulted in incomplete data sets.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 70 | 70
units on a scale
  Baseline | 94.7 (6.8) | 91.9 (9.5)
  1 week: number analyzed (Participants) | 70 | 69
  1 week | 93.4 (7.9) | 88.4 (12.4)

6. Secondary Outcome: Horizontal Centration
Description: Lens fit, horizontal centration will be assessed for senofilcon A and stenfilcon A at baseline for the following regions: extremely nasal, slightly nasal, optimum, slightly temporal, extremely nasal
Time Frame: Baseline
Measure: Number; unit: percentage of subjects
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 70 | 70
percentage of subjects
  Extremely nasal | 0 | 0
  Slightly nasal | 3 | 6
  Optimum | 61 | 73
  Slightly temporal | 36 | 21
  Extremely temporal | 0 | 0

7. Secondary Outcome: Horizontal Centration
Description: Lens fit, horizontal centration, will be assessed for senofilcon A and stenfilcon A at 1 week for the following regions: extremely nasal, slightly nasal, optimum, slightly temporal, extremely nasal
Time Frame: 1 Week
Population: A protocol deviation occurred for 2 participants and therefore resulted in incomplete data sets.
Measure: Number; unit: percentage of subjects
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 69 | 69
percentage of subjects
  Extremely nasal | 0.0 | 0.0
  Slightly nasal | 1.4 | 7.0
  Optimum | 72.5 | 70.0
  Slightly temporal | 26.1 | 23.0
  Extremely temporal | 0.0 | 0.0

8. Secondary Outcome: Vertical Centration
Description: Lens fit, vertical centration, will be assessed for senofilcon A and stenfilcon A at baseline for the following regions: extremely nasal, slightly nasal, optimum, slightly temporal, extremely nasal
Time Frame: Baseline
Measure: Number; unit: percentage of subjects
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 70 | 70
percentage of subjects
  Extremely nasal | 0.0 | 0.0
  Slightly nasal | 17.0 | 15.7
  Optimum | 64.0 | 65.7
  Slightly temporal | 19.0 | 18.6
  Extremely temporal | 0.0 | 0.0

9. Secondary Outcome: Vertical Centration
Description: Lens fit, vertical centration, will be assessed for senofilcon A and stenfilcon A at 1 week for the following regions: extremely nasal, slightly nasal, optimum, slightly temporal, extremely nasal
Time Frame: 1 Week
Population: A protocol deviation occurred for 2 participants and therefore resulted in incomplete data sets.
Measure: Number; unit: percentage of subjects
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 69 | 69
percentage of subjects
  Extremely nasal | 0.0 | 0.0
  Slightly nasal | 20.3 | 23.0
  Optimum | 65.2 | 65.0
  Slightly temporal | 14.5 | 12.0
  Extremely temporal | 0.0 | 0.0

10. Secondary Outcome: Lens Movement
Description: Lens movement assessed for stenfilcon A and senofilcon A at baseline using the following evaluations: extremely inadequate, slightly inadequate, optimum, slightly excessive, extremely excessive.
Time Frame: Baseline
Measure: Number; unit: percentage of subjects
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 70 | 70
percentage of subjects
  Extremely inadequate | 0 | 0
  Slightly inadequate | 29 | 3
  Optimum | 67 | 64
  Slightly excessive | 4 | 33
  Extremely excessive | 0 | 0

11. Secondary Outcome: Lens Movement
Description: Lens movement assessed for stenfilcon A and senofilcon A at 1 week using the following evaluations: extremely inadequate, slightly inadequate, optimum, slightly excessive, extremely excessive.
Time Frame: 1 Week
Population: A protocol deviation occurred for 2 participants and therefore resulted in incomplete data sets.
Measure: Number; unit: percentage of subjects
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 69 | 69
percentage of subjects
  Extremely inadequate | 0 | 0
  Slightly inadequate | 42 | 7
  Optimum | 57 | 65
  Slightly excessive | 1 | 28
  Extremely excessive | 0 | 0

12. Secondary Outcome: Visual Acuity
Description: Measurement of visual acuity (VA) for senofilcon A and stenfilcon A assessed at baseline and 1 week using logMAR VA chart.
Time Frame: Baseline and 1 week
Population: Protocol deviations occurred and therefore resulted in incomplete data sets.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 70 | 70
LogMAR
  Baseline: High Contrast | -0.14 (0.07) | -0.11 (0.08)
  Baseline: Low Contrast | 0.12 (0.10) | 0.16 (0.10)
  1 week: High Contrast: number analyzed (Participants) | 69 | 69
  1 week: High Contrast | -0.13 (0.07) | -0.10 (0.09)
  1 week: Low Contrast: number analyzed (Participants) | 69 | 69
  1 week: Low Contrast | 0.13 (0.09) | 0.17 (0.09)

13. Secondary Outcome: Lens Surface - Deposition
Description: Lens surface for senofilcon A and stenfilcon A is assessed at baseline. Grades 0-4, 0=normal, 1=trace, 2=mild, 3=moderate, 4=severe
Time Frame: Baseline
Measure: Number; unit: percentage of subjects
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 70 | 70
percentage of subjects
  Normal | 94 | 97
  Trace | 6 | 3
  Mild | 0 | 0
  Moderate | 0 | 0
  Severe | 0 | 0

14. Secondary Outcome: Lens Surface - Deposition
Description: Lens surface for senofilcon A and stenfilcon A is assessed at 1 week. Grades 0-4, 0=normal, 1=trace, 2=mild, 3=moderate, 4=severe
Time Frame: 1 week
Population: A protocol deviation occurred for 2 participants and therefore resulted in incomplete data sets.
Measure: Number; unit: percentage of subjects
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 69 | 69
percentage of subjects
  Normal | 91.3 | 99.0
  Trace | 7.2 | 1.0
  Mild | 1.4 | 0.0
  Moderate | 0.0 | 0.0
  Severe | 0.0 | 0.0

15. Secondary Outcome: Lens Surface - Debris
Description: Lens debris for senofilcon A and stenfilcon A is assessed at baseline. Grades 0-4, 0=normal, 1=trace, 2=mild, 3=moderate, 4=severe
Time Frame: Baseline
Measure: Number; unit: percentage of subjects
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 70 | 70
percentage of subjects
  Normal | 82.9 | 93.0
  Trace | 14.3 | 7.0
  Mild | 1.4 | 0.0
  Moderate | 1.4 | 0.0
  Severe | 0.0 | 0.0

16. Secondary Outcome: Lens Surface - Debris
Description: Lens debris for senofilcon A and stenfilcon A is assessed at 1 week. Grades 0-4, 0=normal, 1=trace, 2=mild, 3=moderate, 4=severe
Time Frame: 1 week
Population: A protocol deviation occurred for 2 participants and therefore resulted in incomplete data sets.
Measure: Number; unit: percentage of subjects
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 69 | 69
percentage of subjects
  Normal | 84.1 | 96.0
  Trace | 14.5 | 4.0
  Mild | 1.4 | 0.0
  Moderate | 0.0 | 0.0
  Severe | 0.0 | 0.0

17. Secondary Outcome: Lens Surface - Wettability
Description: Lens wettability for senofilcon A and stenfilcon A is assessed at baseline. Grades 0-4, 0=normal, 1=trace, 2=mild, 3=moderate, 4=severe
Time Frame: Baseline
Measure: Number; unit: percentage of subjects
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 70 | 70
percentage of subjects
  Normal | 79 | 86
  Trace | 20 | 11
  Mild | 1 | 3
  Moderate | 0 | 0
  Severe | 0 | 0

18. Secondary Outcome: Lens Surface - Wettability
Description: Lens wettability for senofilcon A and stenfilcon A is assessed at 1 week. Grades 0-4, 0=normal, 1=trace, 2=mild, 3=moderate, 4=severe
Time Frame: 1 week
Population: A protocol deviation occurred for 2 participants and therefore resulted in incomplete data sets.
Measure: Number; unit: percentage of subjects
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 69 | 69
percentage of subjects
  Normal | 81.2 | 71.0
  Trace | 15.9 | 25.0
  Mild | 1.4 | 4.0
  Moderate | 1.4 | 0.0
  Severe | 0.0 | 0.0

ADVERSE EVENTS:
Arm/Group | Senofilcon A | Stenfilcon A
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other